CLINICAL TRIAL: NCT05285800
Title: To Determine the Effectiveness of Saddle Block vs Spinal Anesthesia in TURP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Wajid Iqbal, Resident medical officer, Anesthesiology, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W0333
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Haemodynamic Instability

STUDY DESIGN:
Intervention Model Description: In Both the groups after injecting 0.5% hyperbaric Bupivacaine intrathecally the outcomes are monitored and compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saddle group (Experimental): After administration of 12mg of 0.5 % Hyperbaric Bupivacaine intrathecally, Patient is advised to remain in Sitting position for the next 5minutes and then take supine position
  Interventions: Drug: 0.5% Hyperbaric Bupivacaine
- Spinal group (Active Comparator): After administration of 12mg of 0.5% Hyperbaric Bupivacaine intrathecally, Patient is advised to take Supine position immediately.
  Interventions: Drug: 0.5% Hyperbaric Bupivacaine

INTERVENTIONS:
Drug: 0.5% Hyperbaric Bupivacaine — In both groups 0.5% Hyperbaric Bupivacaine is given intrathecally and then saddle group is advised to stay in sitting position for next 5minutes so that drug can block only lower segments of nerves, Lumber 5th to Sacral dermatomes level. The spinal group is advised to take supine position immediately so that drug distribution be uniform uptill T10 level of spinal dermatome. Then outcomes regarding haemodynamic status and vasopressor usage are recorded
  Other Names: Hyperbaric Bupivacaine

SUMMARY:
To determine the effectiveness of saddle block vs spinal anesthesia in TURP.

DETAILED DESCRIPTION:
This study is being conducted to determine the effectiveness of saddle block vs spinal anesthesia in terms of haemodynamic stability and Vasopressor usage.

ELIGIBILITY:
Inclusion Criteria:

* Patient with absolute contraindication of general anaesthsia
* Patients who gave consent and willing to be included in study
* Patient's having age range between 45 years to 65years
* Well controlled diabetes and hypertension
* ASA grade I & II

Exclusion Criteria:

* Patients with absolute contraindications of regional anesthesia,
* Deformity of vertebral column,
* Thyroid disorder,
* Psychiatric illness,
* Neurological diseases,
* Alcohol addiction,
* Smoking,
* Ischemic heart diseases and
* Not willing to participate

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
Haemodynamic status | Haemodynamic status checked from 0minutes ( as the patient takes supine position) for every 5minutes interval till the end of surgery.
  Haemodynamic status includes pulse rate, systolic blood pressure, diastolic blood pressure, mean arterial pressure and oxygen saturation.
  Pulse rate ranges between 60-100 beats/ minute. Pulse above 100 is called tachycardia and below 60 is called bradycardia Systolic blood pressure more than 140mmhg is called systolic hypertension and lower than 90mmhg is known as systolic hypotension.
  Diastolic blood pressure more than 90mmhg is called diastolic hypertension and lower than 60mmhg is called diastolic hypotension.
  Mean arterial pressure ranges between 70-110. More than 110 labeled as hypertension and below 70 means hypotension.
  Spo2 level below 94% is labeled as hypoxia.
Vasopressor usage | Blood pressure is taken from 0minute (as the patient takes supine position) at every ⁵minutes interval till the end of surgery
  The main side effect of intrathecal 0.5 % hyperbaric Bupivacaine is hypotension. That is countered by using vasopressor drug e.g inj. Ephedrine. Critically low blood pressure e.g systolic bp below 90mmhg, diastole c blood pressure below 60mmh and MAP below 60 is an indication for vasopressor introduction.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Wajid Iqbal, MBBS, MCPS, Principal Investigator — Hamdard University
Locations (1):
- Dr. Muhammad Wajid Iqbal, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only the study protocol and outcome data will be shared with other researchers in private if the need